CLINICAL TRIAL: NCT04021108
Title: Phase II Study of Short Course FOLFOX Chemotherapy With Either Nivolumab or Nivolumab + Radiation in the First Line Treatment of Metastatic or Unresectable Gastroesophageal Cancers (BMS Protocol CA209-76L)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1812019872
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gastroesophageal Adenocarcinoma
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Other): Subjects will receive standard dose FOLFOX plus nivolumab 240mg IV every 2 weeks for 2 months. If you are responding to treatment, you will receive FOLFOX plus nivolumab for one additional month and then you will be randomized to Cohort 1 or Cohort 2.
  Subjects in Cohort 1 will receive Nivolumab alone (every 2 weeks for two doses, and then every 4 weeks)
  Interventions: Drug: Nivolumab 240 MG
- Cohort 2 (Experimental): Subjects will receive standard dose FOLFOX plus nivolumab 240mg IV every 2 weeks for 2 months. If you are responding to treatment, you will receive FOLFOX plus nivolumab for one additional month and then you will be randomized to Cohort 1 or Cohort 2.
  Subjects in Cohort 2 will receive Nivolumab (every 2 weeks for two doses, and then every 4 weeks) plus radiation therapy (total 5 sessions)
  Interventions: Drug: Nivolumab 240 MG

INTERVENTIONS:
Drug: Nivolumab 240 MG — Nivolumab (OpdivoTM) is a potent and highly selective humanized monoclonal antibody (mAB) designed to block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. Cancer cells are able to send a signal to the PD-1 via the PD-L1 molecule, tricking the T-cell into recognizing the cancer cell as normal. Nivolumab is designed to disrupt that signal and expose the cancer cell to the immune system. Nivolumab is given intravenously over a 60-minute period, usually every two weeks.

SUMMARY:
This is a randomized phase II study examining nivolumab alone versus radiation therapy with nivolumab in subjects who did not have disease progression to initial therapy with the combination of FOLFOX and Nivolumab.

DETAILED DESCRIPTION:
This is a randomized phase II study examining nivolumab alone versus radiation therapy with nivolumab in subjects who did not have disease progression to initial therapy with the combination of FOLFOX and Nivolumab. Subjects with advanced unresectable or metastatic gastroesophageal adenocarcinoma are eligible. All subjects will receive FOLFOX + nivolumab therapy. Subjects who demonstrate at least stable disease, as per RECIST 1.1, on their first imaging assessment at two months will receive one additional month of FOLFOX + nivolumab (3 months total), and then will be randomly assigned at a 1:1 ratio to receive either nivolumab alone or nivolumab plus radiation therapy. Radiation therapy fields and technique will be approved by central review. Radiation will be planned at 4Gy x 5 doses (20 Gy total), given concurrently with nivolumab. After 4 months of therapy, patients who remain on study will receive nivolumab 480 mg every 4 weeks. Subjects will be on study (intervention + follow-up) for approximately 24 months. The projected end date of the study, including data analysis, is February 2026.

ELIGIBILITY:
Inclusion Criteria

* Subjects with a diagnosis of advanced unresectable or metastatic gastroesophageal adenocarcinoma (eg. gastric, gastroesophageal junction, and esophageal adenocarcinoma)
* Be willing and able to provide written informed consent/assent for the trial
* Age > 18 years
* ECOG performance status ≤ 1
* Absolute neutrophil count ≥ 1,500/mL
* Platelets ≥ 100,000/mL
* Total bilirubin ≤ 1.5x upper limits of normal, unless the patient has known Gilbert's disease.
* AST/ALT ≤ 2.5 upper limits of normal, or < 5x ULN for subjects with liver metastases
* Creatinine ≤ 1.5 mg/dl. If Creatinine > 1.5 mg/dl, creatinine clearance > 60 ml/min
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 28 days prior to initiation of treatment on Day 1.
* For all males and females of childbearing potential, they should be agreeable to use an adequate method of contraception or birth control. For females of child bearing potential, a negative pregnancy test within 7 days of start of study drug is required

Exclusion Criteria

* Prior cytotoxic therapy for metastatic or incurable disease.
* Patients may have had prior therapy with curative intent for localized disease, if their recurrence or disease progression was more than six months from completing prior therapy.
* HER2 positive adenocarcinoma
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Known history of active TB (Bacillus Tuberculosis)
* Known additional malignancy that is active. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Previous invasive malignancy treated with curative intent less than 3 years from time of registration. Exceptions include prostate cancer or basal cell skin cancer.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with 12-month progression free survival | 12 months
  This will be measured by number of patients without disease progression at 12 months in the two study arms (patients who receive nivolumab with radiation and those who receive nivolumab alone)

SECONDARY OUTCOMES:
Number of subjects who receive short course chemotherapy with immunotherapy that achieve 12-month progression free survival | 12 months
  This will be measured by the number of patients without disease progression at 12 months in all enrolled patients.
Overall Survival, as measured by the rate of survival in patients | 2 year
  In both study arms, and in all patients together, we will examine the rate of survival in patients over time from registration through their treatment
Occurrence of Significant Toxicity, as measured by Number of Grade 3 and Grade 4 Adverse Events (Combined) Attributable to Immunotherapy | 2 year
  We will measure the rate of grade 3 or 4 adverse events attributable to immunotherapy in both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Roswell Park Cancer Center, Buffalo, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No